CLINICAL TRIAL: NCT03089346
Title: Assessment of Bronchial Thickness Using MRI in Asthma
Acronym: ASTHMAGRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX2016/13
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: Imaging; Bronchial Remodeling
MeSH Terms: conditions — Asthma | interventions — Magnetic Resonance Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asthma (Other): Patients with diagnosis of asthma according to 2016 "Global Strategy for Asthma Management and Prevention (GINA)" definition
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI) with Ultrashort Echo Time (UTE); Diagnostic Test: Computed tomography (CT)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) with Ultrashort Echo Time (UTE) — Magnetic Resonance Imaging (MRI) with Ultrashort Echo Time (UTE) pulse sequences on a 1.5T magnet (Avanto dot, Siemens) with 3D reconstruction of the bronchial tree using Neko-MR software in asthma in order to assess bronchial thickness.
Diagnostic Test: Computed tomography (CT) — Computed tomography (CT) on a Definition 64 (Siemens) with 3D reconstruction of the bronchial tree using Neko-3D software in asthma in order to assess bronchial thickness.

SUMMARY:
Bronchial remodeling is a major pathological feature of asthma. Non-invasive assessment of this bronchial remodeling is a crucial issue for asthma patients' follow-up. Currently, computed tomography (CT) is the method of reference to evaluate and quantify bronchial thickness but it remains unable to differentiate bronchial inflammation from remodelling and is a radiation-based technique. Magnetic Resonance Imaging (MRI) with Ultrashort Echo Time (UTE) pulse sequences is a promising non-ionizing alternative for lung imaging. Our objective is to evaluate bronchial thickness in asthma patients using CT and MRI-UTE, and to test the agreement between both techniques.

DETAILED DESCRIPTION:
Asthma is a major public health problem, pathologically characterized by bronchial remodeling that leads to thickening of the bronchial wall. Computed tomography (CT) is the method of reference to quantify bronchial thickness but involves ionizing radiation, thus limiting the possibility of frequent and long-term follow-up. Magnetic Resonance Imaging (MRI) is a non-ionizing 3D imaging technique. However, lung MRI is technically challenging and is not currently used in routine practice. Indeed, both low proton density and susceptibility effects lead to a very low signal intensity derived from lung parenchyma. Recently, pulse sequences with Ultrashort Echo Time (UTE) have been implemented by the use of half radio-frequency excitations and radial projection reconstruction. These UTE sequences make it theoretically possible to retrieve more signals from the lung parenchyma. We aim at using 3D T1-weighted UTE pulse sequences on a 1.5T magnet (Avanto dot, Siemens) in asthma in order to assess bronchial thickness. Thirty patients with asthma including 10 patients with severe asthma will be enrolled in this study. All participants will benefit from CT and MRI. Our strategy will consist in quantifying bronchial thickness using MRI and CT in those patients, testing for correlations between MRI and CT measurements and assessing the reproducibility of bronchial thickness assessment using MRI. Our objective is to demonstrate that MRI-UTE pulse sequence at 1.5T is accurate and reproducible in evaluating and quantifying bronchial thickness.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged more than 18 years.
* Patients with diagnosis of asthma according to 2016 "Global Strategy for Asthma Management and Prevention (GINA)" definition
* Pulmonary Function Testings (PFTs) should be available within a maximum of 30 days before inclusion.
* With a written informed consent.

Exclusion Criteria:

* Subjects without any social security or health insurance.
* History of chronic obstructive pulmonary disease, lung fibrosis, pulmonary hypertension, lung cancer or cystic fibrosis.
* Pregnancy or breastfeeding women.
* MRI contraindications: Magnetically activated implanted devices (cardiac pacemakers, insulin pumps, neurostimulators, cochlear implants), metal inside the eye or the brain (aneurysm clip, ocular foreign body), cardiac valvular prosthesis (Starr-Edwards pre-6000), subject with claustrophobia, waistline circumference over 200 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the thickness of bronchial wall by MRI | Day 1
  Measurement of quantify bronchial thickness
Evaluation of the thickness of bronchial wall by CT | Day 1
  Measurement of quantify bronchial thickness

SECONDARY OUTCOMES:
Mesure of Pulmonary function | Day 0
  Pulmonary function test
Asthma severity according to GINA 2016 | Day 0
  Asthma severity according to GINA 2016
Presence of bronchiectasis | Day 0
  Observation on the images
Presence of mucoid impaction | Day 0
  Observation on the images
Presence of nodule | Day 0
  Observation on the images
Presence of focal condensation | Day 0
  Observation on the images

CONTACTS AND LOCATIONS:
Overall Officials: Patrick BERGER, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France

IPD SHARING:
Plan to Share IPD: No